CLINICAL TRIAL: NCT01222403
Title: A Multicenter, Post-marketing Surveillance Study to Monitor the Safety of Novartis Vaccine MF59-adjuvanted Influenza Subunit Vaccine FLUAD® and Sandoz Korea Vaccine MF59-adjuvanted Influenza Subunit Vaccine VANTAFLU® Administered According to the Prescribing Information in Korean Subjects Aged 65 Years or Older at the Time of Vaccination.
Brief Title: A Post-marketing Study to Monitor the Safety of a MF59-adjuvanted Influenza Vaccine Administered in Korean Subjects Aged 65 Years or Older
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70_26
Record Dates: First submitted 2010-10-12; First posted 2010-10-18 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Fluad (Experimental): Subjects aged >65 years received one dose of investigational MF59-adjuvanted trivalent influenza vaccine (aTIV).
  Interventions: Biological: Fluad_MF59-adjuvanted trivalent influenza subunit vaccine
- Vantaflu_aTIV (Experimental): Subjects aged >65 years received one dose of investigational MF59-adjuvanted trivalent influenza vaccine (aTIV).
  Interventions: Biological: Vantaflu_MF59-adjuvanted trivalent influenza subunit vaccine

INTERVENTIONS:
Biological: Fluad_MF59-adjuvanted trivalent influenza subunit vaccine
  Arms: Fluad
Biological: Vantaflu_MF59-adjuvanted trivalent influenza subunit vaccine
  Arms: Vantaflu_aTIV

SUMMARY:
This study will evaluate the safety of an influenza (flu) vaccine in Korean men and women aged 65 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 65 years and above on the day of enrollment, who were eligible for seasonal influenza vaccination.
2. In the judgement of the study doctor are determined to be in reasonable health considering their age and able to comply with all study procedures.

Exclusion Criteria:

1. History of any serious reaction to flu vaccine, or any materials in the vaccine, and to eggs (including ovalbumin) and chicken protein.
2. Receipt of another (inactivated) vaccine within 2 weeks, or receipt of a live vaccine within 4 weeks prior to Study Day 1, or planning to receive some other vaccination before the final study visit (about Day 29 after vaccination).
3. Any condition, which in the opinion of the study doctor, might interfere with the evaluation of the study objective.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 767 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- South Korea (22):
  - KeeTaek Kim internal medicine Clinic, Gimpo-si, Gyeonggi-do
  - Jiguchon internal medicine Clinic, Jeongeup, Jeonrabuk-do
  - 21th Century hana internal medicine clinic, Mokpo, Jeonranam-do
  - JoongAng family medicine Clinic, Suncheon, Jeonranam-do
  - Yonsei Universtity College of Medicine, Sinchon-dong, Seoul
  - Hangajok internal medicine clinic, Daejeon
  - Ju Saengmyeong internal medicine Clinic, Daejeon
  - Daejeon hospital, Daejeon
  - SaeSeoul internal medicine and radiology Clinic, Daejeon
  - SeoIncheon catholic clinic, Incheon
  - TaeIl Jang internal medicine Clinic, Incheon
  - SeokYeon Kim internal medicine clinic, Incheon
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Seoul medical center, Seoul
  - Global care internal medicine clinic, Seoul
  - Yeonsei Koum internal medicine Clinic, Seoul
  - Soon Chun Hyang University Hospital, Seoul
  - Gikim internal medicine clinic, Seoul
  - Lee internal medicine clinic, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 24 study sites in Korea.
Pre-assignment Details: All subjects were included in the trial.
Groups:
- Fluad_aTIV: Subjects aged >65 years received one dose of Fluad_aTIV: investigational MF59-adjuvanted trivalent influenza vaccine.
- Vantaflu_aTIV: Subjects aged >65 years received one dose of Vantaflu_aTIV: investigational MF59-adjuvanted trivalent influenza vaccine.
Period: Overall Study
Arm/Group | Fluad_aTIV | Vantaflu_aTIV
Started | 386 | 381
Completed | 386 | 379
Not Completed | 0 | 2
Not completed — Inappropriate enrollment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluad_aTIV | Vantaflu_aTIV | Total
Number analyzed (Participants) | 386 | 379 | 765
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (6.0) | 73.2 (6.5) | 73.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 225 | 456
  Male | 155 | 154 | 309

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events (AEs) After Vaccination.
Description: The number of subjects reporting any solicited local and systemic AEs, following vaccination with Fluad_aTIV and Vantaflu_aTIV.
Time Frame: Day 1 through Day 4 after vaccination
Population: Analysis was done on safety population ie. all subjects in the exposed set who provided postvaccination safety data.
Measure: Number; unit: participants
Arm/Group | Fluad_aTIV | Vantaflu_aTIV
Number analyzed (Participants) | 386 | 379
participants
  Any Local | 134 | 122
  Any Systemic | 74 | 72
  Erythema (Type I) | 14 | 21
  Erythema (Type II) | 9 | 3
  Induration (Type I) | 8 | 14
  Induration (Type II) | 5 | 0
  Swelling (Type I) | 17 | 25
  Swelling (Type II) | 5 | 3
  Pain at injection site | 119 | 111
  Tenderness at injection site | 107 | 98
  Chills | 17 | 20
  Myalgia | 44 | 43
  Arthralgia | 6 | 27
  Headache | 24 | 22
  Sweating | 8 | 15
  Fatigue | 29 | 31

2. Primary Outcome: Number of Subjects Reporting Unsolicited AEs After Vaccination.
Description: The number of subjects reporting any unsolicited AEs following vaccination with Fluad_aTIV and Vantaflu_aTIV.
Time Frame: Day 1 through Day 28 post vaccination
Population: Analysis was done on safety population.
Measure: Number; unit: participants
Arm/Group | Fluad_aTIV | Vantaflu_aTIV
Number analyzed (Participants) | 386 | 379
participants
  Any AEs | 15 | 18
  Possibly/probably related AEs | 3 | 1

3. Primary Outcome: Number of Subjects Reporting Unsolicited Serious Adverse Events (SAEs) After Vaccination.
Description: The number of subjects reporting any unsolicited AEs, SAEs, AEs leading to withdrawal (WD), AEs of special interest (AESI) following vaccination with Fluad_aTIV and Vantaflu_aTIV.
Time Frame: Day 1 through Day 28 post vaccination
Population: Analysis was done on safety population.
Measure: Number; unit: participants
Arm/Group | Fluad_aTIV | Vantaflu_aTIV
Number analyzed (Participants) | 386 | 379
participants
  SAEs | 0 | 0
  At least possibly related SAEs | 0 | 0
  AEs leading to hospitalization | 0 | 0
  AEs leading to interruption or delay | 0 | 0
  AEs resulting in premature withdrawal | 0 | 0
  Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study (Day 1 through Day 28).
Description: All solicited AEs and unsolicited AEs were collected from Day 1 to Day 4; all unsolicited SAEs, medically attended AEs, AEs leading to withdrawal from the study were collected from Day 1 to Day 28.
Arm/Group | Fluad_aTIV | Vantaflu_aTIV
Serious Adverse Events (participants affected / at risk) | 0/386 | 0/379
Other Adverse Events (participants affected / at risk) | 163/386 | 155/379
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluad_aTIV (N=386) | Vantaflu_aTIV (N=379)
Injection site pain (General disorders) | 131 | 121
Fatigue (General disorders) | 29 | 31
Injection site swelling (General disorders) | 17 | 25
Injection site erythema (General disorders) | 14 | 21
Chills (General disorders) | 17 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 44 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 27
Headache (Nervous system disorders) | 24 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days